CLINICAL TRIAL: NCT01507441
Title: Whole Exon Sequencing of Down Syndrome Acute Myeloid Leukemia
Brief Title: Studying DNA in Samples From Younger Patients With Down Syndrome and Acute Myeloid Leukemia Treated on COG-AAML0431 Clinical Trial
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML12B4; COG-AAML12B4 (Other: Children's Oncology Group); AAML12B4 (Other: Children's Oncology Group); NCI-2012-00108 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood myelodysplastic syndromes; childhood acute myeloid leukemia/other myeloid malignancies; childhood acute megakaryocytic leukemia (M7)
MeSH Terms: conditions — Leukemia | interventions — Chromosome Mapping; Microarray Analysis; Base Sequence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene mapping
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: nucleic acid sequencing
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood, tissue, and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies DNA samples from patients with Down syndrome and acute myeloid leukemia treated on COG-AAML0431 clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify new genetic abnormalities associated with acute myeloid leukemia (AML) in patients with Down syndrome through whole-genome sequencing.

OUTLINE: This is a multicenter study.

Extracted DNA and RNA from cryopreserved specimens are analyzed for genomic sequencing, gene mutation, and microarray analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Down syndrome children diagnosed with acute myeloid leukemia (AML) or myelodysplastic syndromes (MDS)
* Clinical samples from patients enrolled on the Children's Oncology Group (COG) AAML0431 phase III clinical trial, and from the Children's Hospital of Michigan Cell Bank

  * Diagnostic blast samples and matched remission samples

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Down syndrome children diagnosed with acute myeloid leukemia (AML) or myelodysplastic syndromes (MDS).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identification of unique mutations through whole-genome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Taub, MD, Principal Investigator — Children's Hospital of Michigan